CLINICAL TRIAL: NCT04152707
Title: Clinical Evaluation of Splendor X for Hair Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-SPLENDOR X-2019-01
Record Dates: First submitted 2019-11-03; First posted 2019-11-05 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Hair Remval

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Splendor X (Experimental)
  Interventions: Device: Splendor X

INTERVENTIONS:
Device: Splendor X — The Splendor X has two wavelengths in one system: Nd:YAG (1064nm) and Alexandrite (755nm).

SUMMARY:
At least 40 healthy male or female subjects that wish to remove their hair will be enrolled to this study.

Each subject will receive five treatments at 6-8 weeks intervals. Subjects will return for follow-up visits at 3, 6, 9, and 12 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. All skin types: I-VI
3. Male or female
4. Age - 18-50 years of age
5. Having one suitable treatment areas (legs, back, Chest or abdomen) with dark brown or black hair appropriate for hair removal;
6. Interested in laser hair removal treatment for permanent hair reduction in the suitable area
7. Able and willing to comply with the treatment/follow-up schedule and requirements;
8. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Pregnant, expectation of pregnancy, postpartum or nursing (<6 months);
2. Participation in another clinical study
3. Active infections in the treated area;
4. Dysplastic nevi in the treatment area;
5. Tattoos in the treatment area;
6. Current cancer, history of skin cancer or pre-cancerous lesions at the treatment areas;
7. History of keloid scars anywhere on the body or scar formation in the treatment area ; or at risk of Keloid scars
8. Active cold sores, open lacerations or abrasions in the treated area;
9. Herpes simplex in the treatment area
10. Prior skin treatment with laser or other devices on the same treated areas prior to study enrollment or during the course of the study
11. Significant concurrent skin conditions or any inflammatory skin conditions;
12. Chronic or cutaneous viral, fungal, or bacterial diseases;
13. Intense tan, Deep suntan, recent suntan within 2 weeks, sunburn or artificially tanned skin;
14. Use of medications, herbal supplements, perfumes or cosmetics that may affect sensitivity to light or change skin metabolism
15. Skin lesions
16. Bleeding coagulopathies or use of anticoagulants
17. Hormonal disorders that may affect hair growth;
18. Immunosuppressive diseases, including AIDS and HIV infection, or use of immunosuppressive medications; or other auto-immune dsorders.
19. Livedo reticularis;
20. Uncontrolled systemic diseases such as diabetes;
21. Use of Accutane™ (Isotretinoin) within the past 6 month;
22. Erythema ab igne, when identified treatments should be discontinued;
23. Photosensitivity disorder that can be exacerbated by laser or intense light (such as Epilepsy).
24. Poor wound healing;
25. Unable or unlikely to refrain from artificial tanning, including the use of tanning booths, prior (at least 6 week) and during the course of the evaluation;
26. Previous skin procedures on requested treatment area (botox, fillers , peels , lasers etc. )
27. Mechanical or chemical hair removal in the treated area within 6 weeks before the laser treatment
28. Subjects who do not desire permanent hair reduction in the areas to be treated
29. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Hair reduction | 3 months follow up
  change in number of hairs at 3 months following the last treatment as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rohrer, Dr., Principal Investigator — SkinCare Physicians; Anne Chapas, Dr., Principal Investigator — Union Square Laser Dermatology
Locations (2):
- United States (2):
  - SkinCare Physicians, Boston, Massachusetts
  - Union Square Laser Dermatology, New York, New York